CLINICAL TRIAL: NCT00493740
Title: Cephalic Phase of Oncology Patients Before and After Chemotherapy as Compared to Healthy Controls
Acronym: Cephalic chemo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TASMC-07-NV-218-CTIL
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-06

CONDITIONS: Cephalic Phase, Oncology Patients
Keywords: Cephalic phase, oncology patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: chocolate cake

SUMMARY:
The objective of this trial is to examine the cephalic phase insulin response (CPIR) and pancreatic polypeptide (PP) release as indicators of the cephalic phase occurrence and magnitude to palatable food stimulus (chocolate cake) in oncology patients before and after chemotherapy treatment as compared to healthy controls . This may enlighten our understanding of the etiology of taste dysfunction and anorexia during chemotherapy treatments.

DETAILED DESCRIPTION:
Food stimulation of gastric and pancreatic secretion is classically divided into cephalic, gastric and intestinal phases.

Cephalic phase refers to a simultaneous activation of gastrointestinal motility, gastric acid and pancreatic enzyme secretion ,as well as, release of hormones from the endocrine pancreas which occurs through activation of vagal -efferents as a result of food-related sensory stimuli such as taste and smell prior to nutrient absorption and which coincides with a thermogenic response.

Of the cephalic phase secretions, cephalic phase insulin release (CPIR) has received the most attention, but pancreatic polypeptide (PP) and glucagon responses have also been studied. While the magnitude of cephalic phase insulin release is relatively small (25% above baseline), pancreatic polypeptide increases 100% above baseline. The large magnitude of the PP response makes it a sensitive indicator of vagal activation to food stimuli.

In most experiments, subjects are either exposed to visual and olfactory stimulation by seeing and smelling the food stimulus or are required to perform a modified sham-feed, i.e. to taste, chew and then expectorate the food stimulus.

In general, cephalic phase are thought to be preparatory responses before ingestion of food. Because of their small magnitude, the physiological significance of the cephalic phase hormonal responses has been largely discounted. However, there is evidence that experimental prevention of CPIR lead to hyperinsulinemia and hyperglycemia. Therefore, CPIR may contribute to glucose homeostasis /regulation. Moreover CPIR may be an indicator of hunger and could be important for understanding eating disorders.

In parallel with these hormonal secretion ,an increase in energy expenditure has been also observed .This thermogenic response to food is even greater with sham feeding than with normal feeding and is paralleled by changes in RQ showing enhanced carbohydrate oxidation.

Disorders of taste are prevalent symptom in patients undergoing chemotherapy. The literature suggests that 36% to71% of patients report a distressing change in taste which often have a negative impact on quality of life and nutrition. It is unknown whether the cephalic phase of oncology patients may also be disturbed.

ELIGIBILITY:
Subjects:

40 oncology patients of the following 3 subgroups will be recruited from the oncology out-patient department;

1. . 10 un-operated sigmoid rectal cancer patients (i.e. metastatic stage) before treatment and after 2 months of treatments with Avastin + 5FU + CPT only.
2. . 10 un-operated sigmoid rectal cancer patients (i.e. metastatic stage) before treatment and after 2 months of treatments with Oxaliplatin + 5FU + Avastin.
3. . 10 operated sigmoid rectal cancer patients before the operation and 2 months after the operation.
4. . 10 control healthy subjects, age, sex and BMI matched.

Inclusion\Exclusion criteria:

Non diabetic and non-pregnant oncology patients above 18 years of age who are not on steroids and medications which can stimulate appetite.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-07; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
VAS, EDI, Blood test for glucose, insulin, PP, shame feed procedure | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, Prof., Principal Investigator — TASMC
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel